CLINICAL TRIAL: NCT03246607
Title: Investigation of Venous and Cerebral Extracellular Glucose Concentration Relationship Using Continuous Microdialysis, in Acquired Brain Injury in Neurocritical Care, With External Validation of Venous Microdialysis System
Brief Title: Venous and Cerebral Glucose Microdialysis in Neurocritical Care: Validation & Correlation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr Andrew Stevens (Other)
Collaborators: Probe Scientific Limited (Industry)
Responsible Party: Sponsor-Investigator, Dr Andrew Stevens, Academic Foundation Doctor, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: NCCUGLUC/8817
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Traumatic Brain Injury; Acquired Brain Injury; Intracerebral Hemorrhage; Subarachnoid Hemorrhage; Ischemic Stroke
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Cerebral Hemorrhage; Subarachnoid Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monitoring with MicroEye & ContinuMon: 72 hour study interval with monitoring using intravascular glucose monitoring system alongside routine clinical care.
  Interventions: Device: MicroEye & ContinuMon

INTERVENTIONS:
Device: MicroEye & ContinuMon — Continuous intravascular glucose monitoring using MicroEye/ContinuMon system, peripherally inserted via a peripheral venous catheter.

SUMMARY:
This study evaluates the validity of an intravascular continuous glucose monitoring microdialysis probe, and compares the values to routinely inserted cerebral glucose microdialysis to evaluate the hypothesised relationship between intracranial and intravascular glucose levels.

DETAILED DESCRIPTION:
All recruited patients will in any case have probes inserted in theatre for brain tissue glucose monitoring as a part of their standard clinical care. Probes will be allowed to stabilize following insertion as is standard clinical practice. A peripheral venous catheter will be inserted by the study team to allow introduction of the intravascular microdialysis probe. This will be attached to a regular infusion pump set at 3ml/hr and normal saline, to produce the microdialysate. The efflux of microdialysate will be connected to the biosensor, and once passed over the biosensor the subsequent dialysate will be destroyed. A risk assessment will be made on the basis of the patient's coagulation status and concurrent venous thromboembolism prophylaxis, and if necessary, low dose low molecular weight heparin will be included in the saline infusion to ameliorate risk of local thrombosis in the device. This has a local effect only and does not produce systemic anticoagulation.

After a brief period of probe stabilisation, 2 ml of blood will be withdrawn for blood gas analysis (including glucose), and the probe readings will be calibrated against this value. Subsequent calibration will take place 6 hours later, and then at 12 hourly intervals. A maximum total of 30ml of blood will be required for each patient for blood oxygen content analysis. Clinically necessitated blood sampling for blood gases will continue, and these values will be collected post-hoc from our E-hospital clinical records system.

Further data will be collected post-hoc via e-Hospital clinical records system, including: routinely recorded measures of cerebral extracellular fluid glucose concentration, physiological parameters (central venous pressure, mean arterial pressure, intracranial pressure etc), timing and detail of interventions as determined appropriate by routine clinical decision making.

The study will terminate at 72 hours, whereupon the device will be detached and the peripheral venous catheter will be removed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16 and over
2. New episode of acquired brain injury, of any form to include haemorrhage, trauma, infarction
3. Their condition necessitates admission to and care on neurocritical care
4. Their condition necessitates intracerebral microdialysis probe insertion
5. Their condition necessitates arterial line insertion/central venous access and regular/venous blood gas sampling.

Exclusion Criteria:

1. Refusal or withdrawal of consultee agreement and any known patient wishes precluding inclusion.
2. Pregnancy.
3. Peripheral venous cannulation clinically contraindicated.
4. Patients already enrolled in three or more other research studies.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are admitted to the Neurocritical Care Unit with a severe acquired brain injury
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-26 (Estimated); Primary Completion 2020-08-02 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Continuously measured intravascular glucose concentration | 72 hours
  Study inserted microdialysis catheter for collection of data on the concentration of glucose in this space.

SECONDARY OUTCOMES:
Intermittently measured intravascular glucose concentration | 72 hours
  Routinely collected data on the concentration of glucose in this space at specific time points.
Cerebral extracellular fluid glucose concentration | 72 hours
  Routinely inserted microdialysis catheter for collection of data on the concentration of glucose in this space.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Ercole, PhD, Principal Investigator — Lecturer and Consultant Anaesthetist; Peter Hutchinson, PhD, Principal Investigator — NIHR Research Professor at the Department of Clinical Neurosciences
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No